CLINICAL TRIAL: NCT00042770
Title: Phase III Comparison of Catheter Based Therapy of Pleural Effusions in Cancer Patients (Optimal Pleural Effusion Control, OPEC)
Brief Title: Standard Chest Tube Compared With a Small Catheter in Treating Malignant Pleural Effusion in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30102; U10CA076001 (NIH); CALGB-30102; CDR0000069451 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Cancer; Pulmonary Complications
Keywords: malignant pleural effusion; pulmonary complications
MeSH Terms: conditions — Neoplasm Metastasis; Pleural Effusion, Malignant | interventions — Talc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo placement of a standard pleural chest tube. Within 36 hours of chest tube placement, patients undergo pleurodesis comprising intrapleural administration of talc slurry once followed by clamping of the chest tube for 2 hours while different patient positions are used to distribute the talc. The chest tube is then unclamped to allow continuous drainage. When the chest tube drainage is less than 150 mL over 24 hours, pleurodesis is assumed and the chest tube is removed.
  Interventions: Other: talc
- Arm II (Experimental): Patients undergo pleurodesis comprising placement of a small (PleurX) catheter followed by pleural drainage for up to 90 minutes once daily. When the catheter drainage is less than 30 mL per day for 3 consecutive days, pleurodesis is assumed and the catheter is removed.
  Interventions: Procedure: dyspnea management

INTERVENTIONS:
Other: talc — Given intrapleurally
  Arms: Arm I
Procedure: dyspnea management — No talc
  Arms: Arm II

SUMMARY:
RATIONALE: It is not yet known whether pleurodesis using a chest tube with infusions of talc is more effective in improving quality of life than pleurodesis using a small catheter in treating malignant pleural effusion.

PURPOSE: Randomized phase III trial to compare the effectiveness of a chest tube and talc with that of a small catheter in treating malignant pleural effusion in patients who have cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the success rate in patients with cancer who undergo pleurodesis using a standard chest tube with talc slurry vs a small (PleurX) catheter for the treatment of a symptomatic unilateral malignant pleural effusion.
* Compare the 30-day effusion control rate in patients treated with these procedures.
* Compare quality of life in these patients at 7-14 and 30-37 days after treatment with these procedures.
* Compare patient acceptance and satisfaction after treatment with these procedures.
* Compare the level of symptoms and dyspnea experienced by patients treated with these procedures.
* Compare the types, causes, and rates of early technical failures of these procedures in these patients.
* Compare the 30-day effusion recurrences in patients treated with these procedures.
* Compare the 60-day durability of pleurodesis in patients treated with these procedures.
* Compare the mortality, morbidity, and common surgical complications in patients treated with these procedures.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to inpatient status (yes vs no), disease type (breast vs lung vs other), and concurrent systemic chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo placement of a standard pleural chest tube. Within 36 hours of chest tube placement, patients undergo pleurodesis comprising intrapleural administration of talc slurry once followed by clamping of the chest tube for 2 hours while different patient positions are used to distribute the talc. The chest tube is then unclamped to allow continuous drainage. When the chest tube drainage is less than 150 mL over 24 hours, pleurodesis is assumed and the chest tube is removed.
* Arm II: Patients undergo pleurodesis comprising placement of a small (PleurX) catheter followed by pleural drainage for up to 90 minutes once daily. When the catheter drainage is less than 30 mL per day for 3 consecutive days, pleurodesis is assumed and the catheter is removed.

Quality of life and dyspnea are assessed at baseline and then at 7-14 and 30-37 days after treatment.

Patients are followed at 30 and 60 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologic evidence of a unilateral malignant pleural effusion requiring sclerosis or ongoing drainage because it is symptomatic (dyspnea and/or progressive fatigue)

  * An asymptomatic patient is eligible if the patient underwent a prior thoracentesis within the past 2 weeks and was symptomatic before the procedure
  * No bilateral effusions by plain chest x-ray
* Histologically or cytologically confirmed solid tumor or hematologic malignancy

  * Histologic confirmation of malignant cells in pleural fluid is not required
* Pleural spaces must be naive to pleurodesis attempts

  * No prior intrapleural therapy (defined as a chest tube in place or placed to drain an effusion, prior surgical pleurectomy, or any prior chemical or mechanical pleurodesis on the ipsilateral side)

    * Placement of a small interventional radiology catheter for temporary drainage is not considered intrapleural therapy as long as no sclerosant medication was given and it has not been in place longer than 10 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* CTC 0-2

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Pulmonary

* No active pleural infection

Other

* No allergy to talc
* No surgical contraindication to talc usage
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy

* Concurrent systemic chemotherapy allowed

Radiotherapy

* Concurrent palliative radiotherapy to a symptomatic lesion allowed except to the treated hemithorax within 30 days of the drainage procedure

Surgery

* See Disease Characteristics
* Prior thoracotomies without specific pleural ablation (including lobectomy but not pneumonectomy) allowed
* Prior needle-based diagnostic interventions (fine-needle aspiration, small bore catheter drainage of less than 10 days, or thoracentesis) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-05; Primary Completion 2005-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Effusion control | 30 days

SECONDARY OUTCOMES:
Quality of Life | 7-14 days and 30-37 days

CONTACTS AND LOCATIONS:
Overall Officials: Todd Demmy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Providence Saint Joseph Medical Center - Burbank, Burbank, California, United States